CLINICAL TRIAL: NCT01594372
Title: Randomized Trial Comparing Vaginal Hysterectomy to Laparoscopic Supracervical Hysterectomy With Vault Suspension for Symptomatic Uterine Prolapse
Brief Title: Comparison of Laparoscopic to Vaginal Surgical Repair for Uterine Prolapse
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Laproscopic procedure not offered at this time; will not be offered for the foreseeable, thus we are unable to randomize participants between the two arms.
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Vatche Arakel Minassian, Director of Urogynecology, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VM-2012-01
Record Dates: First submitted 2012-05-04; First posted 2012-05-09 (Estimated); Last update posted 2022-03-04 (Actual); Status verified 2022-03

CONDITIONS: Uterine Prolapse
Keywords: Uterine Prolapse; Laparoscopy; Hysterectomy, vaginal
MeSH Terms: conditions — Uterine Prolapse | interventions — Hysterectomy, Vaginal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Laparoscopic Repair (Active Comparator): Laparoscopic supracervical hysterectomy with sacropexy
  Interventions: Procedure: Laparoscopic supracervical hysterectomy with sacropexy
- Vaginal Repair (Active Comparator): Vaginal hysterectomy with uterosacral colposuspension
  Interventions: Procedure: Vaginal hysterectomy with uterosacral colposuspension

INTERVENTIONS:
Procedure: Laparoscopic supracervical hysterectomy with sacropexy — Will involve laparoscopic entry to the abdomen to remove the uterus and suspension of the cervix and vaginal cuff to the sacrum with mesh. We will allow surgeons to conduct the surgery as they have perfected it
  Arms: Laparoscopic Repair
Procedure: Vaginal hysterectomy with uterosacral colposuspension — Will involve removing the uterus vaginally followed by suspending the vaginal cuff to the high (proximal) uterosacral ligaments bilaterally restoring the vagina to its normal axis.
  Arms: Vaginal Repair

SUMMARY:
Investigators intend to conduct a prospective randomized trial to compare vaginal hysterectomy with uterosacral colposuspension to laparoscopic supracervical hysterectomy with sacrocervicopexy. Both surgeries are minimally-invasive surgical standards of care for uterine prolapse repair. Nobody knows if one procedure is superior to the other, as they have not been compared directly. The investigators hypothesize that there is no difference in objective, subjective, or cost-effectiveness between the two procedures for up to two years after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary symptomatic uterine prolapse
* ≥ 18 years of age
* Considering pelvic reconstructive surgery

Exclusion Criteria:

* Unwillingness to be randomized to one of two surgical approaches
* Pregnant or planning to maintain their future fertility
* Unable to have general anesthesia
* Currently undergoing chemotherapy OR has current or history of pelvic radiation
* Previous adverse reaction to synthetic mesh
* Recent history of abnormal paps (past 10 years)
* Cervical or uterine cancers
* Previous hysterectomy
* Previous central vault or uterine prolapse repair
* Uterus ≥ 14 weeks size
* Uterine cancer
* History of significant pelvic adhesive disease
* Elongated cervix (length D to C > 6cm)
* Fibroid ≥ 7cm
* Post menopausal with enlarged uterus

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2013-01; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Whether or not POPQ points AA, BA, Ap, or Bp are at less than 0 cm from the hymen OR whether point C descends less than 1/3 of the total vaginal length (TVL) | 24 months
Absence of re-treatment for prolapse at 2 years | 24 months
A negative response to "Do you usually have a bulge or something falling out that you can see or feel in the vaginal area?" | 24 months
  This is a question from the standardized questionnaire called Pelvic Floor Discomfort Inventory (PFDI).

SECONDARY OUTCOMES:
Changes in POPQ measurements | baseline, 6 week, and 3, 12, and 24 months
Changes in Patient-reported quality of life scores from the EQ-5D, PFDI, PFIQ, SF-12, Standard Gamble Interview, Pain Scale and Activity Assessment | baseline, 3, 12, and 24 months
  EQ-5D assesses a patient's health that day PFDI- pelvic floor discomfort questions PFIQ - pelvic floor impact on daily activity questions SF-12 - general health/quality of life questions Standard Gamble Interview - an overall general health/quality of life questionnaire
Change in patient reported sexual questionnaire, PISQ | baseline, 3, 12 and 24 months
  PISQ - pelvic organ prolapse/urinary incontinence sexual questionnaire
Frequencies of surgical and post-operative complications | up to 2 years post-operatively
  Complications will be classified and reported, based on severity.

CONTACTS AND LOCATIONS:
Overall Officials: Vatche A Minassian, MD, MPH, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham And Women's Hospital, Boston, Massachusetts, United States